CLINICAL TRIAL: NCT01833780
Title: Effectiveness of Intrapartum Group B Streptococcus (GBS) Polimerase Chain Reaction Reaction (PCR) Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Yuri perlitz, Director, High Risk Unit, Department of OB&GYN, The Baruch Padeh Medical Center, Poriya, The Baruch Padeh Medical Center, Poriya
Other Study IDs: GBS PCR .CTIL
Record Dates: First submitted 2013-04-08; First posted 2013-04-17 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: GBS
Keywords: carriage status; Culture; PCR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (2):
- GBS carriage status
- GBS status during labor

SUMMARY:
Study hypothesis: Intrapartum polimeraze chain reaction (PCR)of group B streptoccocus (GBS) test is more accurate than Culture of GBS at 35-37 weeks gestation for GBS carriage.

The investigators will compare GBS culture and PCR results taken at 35-37 weeks gestation to intrapartum PCR GBS and GBS cultures status.

The larger perspective of this trial is to check the possibility of replacing the GBS culture screening program at 35-37 weeks gestation with a more accurate examination (PCR), avoiding the changing GBS carriage status from the time of culture at 35-37 weeks to delivery.

ELIGIBILITY:
Inclusion Criteria:

* Unknown GBS pregnant women at 35-37 weeks

Exclusion Criteria:

* Known GBS pregnant women at 35-37 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Unknown GBS pregnant women
Sampling Method: Probability Sample
Dates: Start 2013-05; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Intrapartum GBS carriage staus measured by PCR and culture compared to GBS culture and PCR at 35-37 weeks gestation | One year
  Intrapartum GBS carriage status measured by culture and PCR will be compared to GBS carriage stauts measured by the same tests at 35-37 weeks gestation.